CLINICAL TRIAL: NCT07320586
Title: Clinical Study on the Combination of Carilizumab and Albumin Paclitaxel for Second-line Treatment of Advanced Gastric Cancer Patients Who Have Received/Not Received Immunotherapy in the Past
Brief Title: Carilizumab and Albumin Paclitaxel for Second-line Treatment of Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Tumor Hospital (Other)
Responsible Party: Principal Investigator, Xiuping Ding, Dr, Shandong Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-010
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Second-line Therapy
Keywords: Immune checkpoint inhibitors；; Camrelizumab
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; Taxes; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Subjects with advanced gastric cancer who have been included in first-line treatment and have received systemic chemotherapy in the past.
  Administration method: Camrelizumab 200mg, d1, q3w, Albumin bound paclitaxel 100mg/m2 on days 1 and 8, q3w， Treatment until disease progression, toxicity intolerance, initiation of new anti-tumor therapy, withdrawal of information or researcher's judgment that the subject needs to withdraw from the study treatment. The longest duration of administration for Camrelizumab is 2 years, while the longest duration of treatment for albumin bound paclitaxel is 6-8 cycles.
  Interventions: Drug: Camrelizumab; Drug: Nab paclitaxel
- Group 2 (Experimental): Advanced gastric cancer subjects included in the first-line treatment progression, who have previously received systemic chemotherapy combined with immunotherapy in the first-line treatment Administration method: Camrelizumab 200mg, d1, q3w, Albumin bound paclitaxel 100mg/m2 on days 1 and 8, q3w， Treatment until disease progression, toxicity intolerance, initiation of new anti-tumor therapy, withdrawal of information or researcher's judgment that the subject needs to withdraw from the study treatment. The longest duration of administration for Camrelizumab is 2 years, while the longest duration of treatment for albumin bound paclitaxel is 6-8 cycles.
  Interventions: Drug: Camrelizumab; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg，d1，q3w.Treatment until disease progression, toxicity intolerance, initiation of new anti-tumor therapy, withdrawal of information or researcher's judgment that the subject needs to withdraw from the study treatment. The longest duration of use for Carilizumab is 2 years
Drug: Nab paclitaxel — nab-paclitaxel 100mg/m2 D1、8，q3w， Treatment until disease progression, toxicity intolerance, initiation of new anti-tumor therapy, withdrawal of information or researcher's judgment that the subject needs to withdraw from the study treatment. The longest treatment time for albumin bound paclitaxel is 6-8 cycles.
  Other Names: nab-paclitaxel

SUMMARY:
This study was an open, single center, prospective cohort study design. Subjects with advanced gastric cancer who had received first-line chemotherapy (cohort 1) and systematic chemotherapy combined with immunotherapy (cohort 2) were included in this study. 20 cases were included in each population, and a total of 40 subjects were planned to be included.

DETAILED DESCRIPTION:
1. main research purposes: Objective To observe the objective response rate (ORR) of carrelizumab combined with albumin paclitaxel in the second-line treatment of patients with advanced gastric cancer who previously received or did not receive immunotherapy.
2. secondary research purposes: Objective To observe the progression free survival (PFS), overall survival (OS), disease control rate (DCR) and safety of carrelizumab combined with albumin paclitaxel in the second-line treatment of patients with advanced gastric cancer who received or did not receive immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18 to 75 years old, both male and female are acceptable;
2. Patients with gastric adenocarcinoma or gastroesophageal junction adenocarcinoma diagnosed by histology or cytology;
3. Gastric cancer patients who have previously received first-line systemic chemotherapy (queue 1) or systemic chemotherapy combined with immunotherapy (queue 2) for progression; For intervention group 2, the best response to first-line immunotherapy is CR or PR or SD ≥ 3 months;
4. According to the evaluation criteria for solid tumor efficacy 1.1 (RECIST v1.1), there should be at least one measurable lesion that has not received local treatment such as radiotherapy (lesions located within the previously irradiated area can also be selected as target lesions if progression is confirmed);
5. ECOG score: 0-1 point;
6. Expected survival period ≥ 12 weeks;
7. The main organ functions well and the laboratory test data meets the following standards: (1) Blood routine: absolute neutrophil count ≥ 1.5 × 109/L (or greater than the lower limit of normal laboratory values in the research center), platelet count ≥ 100 × 109/L, hemoglobin ≥ 90g/L; (2) Liver function: serum total bilirubin ≤ 1.5 times the upper limit of the standard value (ULN), AST and ALT ≤ 2.5 times ULN. If the patient has liver metastasis, this standard is ≤ 5 times ULN; (3) Renal function: CrCl ≥ 60 ml/min/1.73 m2 (calculated according to the Cockcroft Gault formula);
8. Female subjects with fertility, as well as male subjects with partners who are fertility women, are required to use a medically approved contraceptive measure (such as intrauterine devices, birth control pills, or condoms) during the study treatment period, at least 6 months after the last use of Carilizumab, and at least 6 months after the last use of chemotherapy;
9. HER2 negative;
10. Voluntarily join this study, sign the informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. History of gastrointestinal perforation and/or fistula within 6 months prior to the first use of medication;
2. There is uncontrollable pleural effusion, pericardial effusion, or peritoneal effusion that requires repeated drainage;
3. History of allergies to monoclonal antibodies, any component of Carilizumab, or albumin bound paclitaxel;
4. Have received any of the following treatments:

   1. Patients who have experienced serious adverse reactions to immunotherapy in the past and are deemed unsuitable for continued use of immunotherapy by the researchers;
   2. Received any other investigational drug within 4 weeks prior to the first use of the investigational drug or had a half-life of no more than 5 from the last investigational drug;
   3. Simultaneously enrolled in another clinical study, unless it is an observational (non interventional) clinical study or an interventional clinical study follow-up;
   4. Received anti-tumor therapy (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, or tumor embolization) within 2 weeks prior to the first use of the investigational drug;
   5. Subjects who need to receive corticosteroids (equivalent to>10mg prednisone per day) within 2 weeks prior to the first use of the study drug. Other special circumstances require communication with the researcher. In the absence of active autoimmune diseases, inhalation or local use of steroids and corticosteroids with a dosage greater than 10mg/day of prednisone efficacy dose are allowed as substitutes for adrenal cortex hormones;
   6. Individuals who have received anti-tumor vaccines or have received live vaccines within 4 weeks prior to the first administration of the study drug;
   7. Having undergone major surgery or suffered severe trauma within 4 weeks prior to the first use of the investigational drug;
   8. Patients who have received previous treatment with paclitaxel drugs;
5. The toxicity of previous anti-tumor treatments has not recovered to ≤ CTCAE 5.0 Grade 1 (excluding hair loss) or the level specified in the inclusion/exclusion criteria;
6. Patients with central nervous system metastases;
7. Active autoimmune diseases, history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to the above diseases or syndromes); Excluding childhood asthma/allergies with vitiligo or those who have already recovered, patients who do not require any intervention in adulthood; Autoimmune mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes with a stable dose of insulin;
8. Have a history of immune deficiency, including HIV test positive, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation and allogeneic bone marrow transplantation, or active hepatitis (hepatitis B reference: HBV DNA test value exceeds 500 IU/ml or 2500 copies/mL);
9. The subject has uncontrolled cardiovascular clinical symptoms or diseases, including but not limited to: (1) NYHA class II or above heart failure; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within one year; (4) Clinically significant supraventricular or ventricular arrhythmias that have not been clinically intervened or are still poorly controlled after clinical intervention;
10. Within 4 weeks prior to the first use of the investigational drug, there has been a severe infection (CTCAE 5.0>grade 2), such as severe pneumonia requiring hospitalization, bacteremia, infection complications, etc; Baseline chest imaging examination suggests the presence of active pulmonary inflammation, symptoms and signs of infection within 2 weeks prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment, except for prophylactic use of antibiotics;
11. History of interstitial lung disease (excluding history of radiation pneumonia and non infectious pneumonia that have not been treated with steroids);
12. Patients with active pulmonary tuberculosis infection found through medical history or CT examination, or patients with a history of active pulmonary tuberculosis infection within the past year before enrollment, or patients with a history of active pulmonary tuberculosis infection more than one year ago but without formal treatment;
13. Diagnosed with any other malignant tumor within 5 years prior to the first use of the investigational drug, except for malignant tumors with low-risk metastasis and mortality risk (5-year survival rate>90%), such as basal cell or squamous cell carcinoma or cervical carcinoma in situ that have been adequately treated;
14. Pregnant or lactating women;
15. According to the researcher's assessment, there may be other factors that could force the subject to terminate the study midway, such as having other serious illnesses (including mental illnesses) that require concurrent treatment, severe abnormal laboratory test values, family or social factors that may affect the subject's safety or the collection of trial data.
16. According to the researcher's assessment, there may be other factors that could force the subject to terminate the study midway, such as having other serious illnesses (including mental illnesses) that require concurrent treatment, severe abnormal laboratory test values, family or social factors that may affect the subject's safety or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
mPFS | [Time Frame: The longest follow-up period from the patient's enrollment to disease progression or death from any cause is 2 years]
  median Progression free survival

SECONDARY OUTCOMES:
mOS | [Time Frame: The longest follow-up period from the patient's enrollment todeath from any cause is 2 years]
  median survival time
DCR | [Time Frame: The longest follow-up period from enrollment to the first efficacy evaluation is 3 months]
  Disease Control Rate
safety：Record the incidence rate of all adverse events | [Time Frame: From enrollment until 90 days after the last dose of medication]
  Record the incidence rate of all adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Zuoxing Niu, Professor, Principal Investigator — Shandong First Medical University Affiliated Cancer Hospital
Locations (1):
- Shandong First Medical University Affiliated Cancer Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided